CLINICAL TRIAL: NCT05196529
Title: Inspiratory Muscle Training in Myalgic Encephalomyelitis/Chronic Fatigue Syndrome (ME/CFS) and COVID-19 Survivors
Brief Title: Inspiratory Muscle Training in ME/CFS and COVID-19 Survivors
Acronym: Inspire ME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: York University (Other)
Responsible Party: Principal Investigator, Heather Edgell, Associate Professor, York University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: SOLVE ME/CFS
Record Dates: First submitted 2022-01-13; First posted 2022-01-19 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Myalgic Encephalomyelitis; Post-acute COVID-19 Syndrome
MeSH Terms: conditions — Fatigue Syndrome, Chronic; Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Intervention Model Description: Three groups (controls, ME/CFS, COVID long-haulers) will all conduct an inspiratory training protocol and cardiovascular and autonomic measures will be measured before and after.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Inspiratory muscle training (Experimental): The 8-week inspiratory muscle training protocol consists of using 80% of maximal inspiratory pressure (determined in lab), 3x per week, 6 sets of 6 repetitions. Each set will be separated by decreasing lengths of time over the 8 weeks starting at a 30 second interim. This totals 36 inhalations 3 times per week. Progress will be determined via weekly phone calls with the participants and progress will also be logged by participants over the 8 weeks.
  Interventions: Other: Inspiratory muscle training

INTERVENTIONS:
Other: Inspiratory muscle training — All participants will undergo inspiratory muscle training.

SUMMARY:
Coronavirus-2019 (COVID-19) is a viral disease leading to respiratory dysfunction, but it may also affect the brain and result in the development of myalgic encephalomyelitis/chronic fatigue syndrome (ME/CFS). This may be the result of the COVID-19 virus infecting regions of the brain responsible for respiratory control. The symptoms of COVID-19 long haulers and ME/CFS may be lessened via an 8-week inspiratory muscle training protocol which is a simple and easy training protocol which can be done at a patient's home.

Thus, this project will investigate changes in the breathing and cardiovascular responses to stimuli in three groups of participants: 1) healthy control individuals; 2) patients diagnosed with ME/CFS (mild to moderate symptoms); and 3) individuals with previous COVID-19 infection with long-haul symptoms lasting for at least 3 months. Participants will 1) breathe hypoxic gas (10% O2) for 5 minutes; 2) breath hypercapnic gas (5% CO2) for 5 minutes; 3) breathe at a rate of 6 breaths per minute for a total of 8 breaths (paced deep breathing); and 4) complete 10 minutes upright tilt (70 degrees head up on a tilt-table). Patients will also complete 2 questionnaires concerning their symptoms and a 15 minute cognitive function test on a lab laptop. This will allow for the assessment of the brain's control over blood pressure and breathing. Participants will also complete a 6-minute walking exercise test at their own speed as a measure of their aerobic fitness. We hypothesize that COVID-19 survivors will have a worse cardiovascular and autonomic response and lower fitness, similar to ME/CFS patients, compared to healthy participants.Further, this will be improved after 8-weeks of inspiratory muscle training. These results may help clinicians recognize ME/CFS symptoms in patients recovering from COVID-19.

DETAILED DESCRIPTION:
Approximately 10 women and 10 men between the ages of 18-65 will be tested in each of 3 groups:

1. Control participants will be free of previously diagnosed cardiovascular, metabolic, autonomic, or respiratory disease.
2. COVID-19 participants will have both an official diagnosis and an official clearance of COVID-19. Patients will have long-haul symptoms for at least 3 months. Patients will be recruited via media, social media and clinical collaborators.
3. ME/CFS participants will be recruited via media, social media and clinical collaborators. Only those with mild to moderate symptoms who can complete a 6 minute walk test will be recruited.

Prospective participants will be patients of the University Health Network (UHN) or Women's College Hospital, community members, friends, family, and co-workers of laboratory staff and students. Patients will be recruited from clinical sites by poster recruitment at collaborative clinics.

Exclusion criteria are severe symptoms of chronic fatigue syndrome, inability to stand on a tilt table, inability to walk for 6 minutes, previous cardiorespiratory disease (except for COVID-19 long-hauler symptoms and chronic fatigue syndrome itself), and inability to understand and read English.

Participants will be recruited via established clinical collaborators, from York University's student and staff population, previously known relationships with the research staff, poster recruitment, and advertisements on social media sites (e.g. York U reddit, Facebook, Instagram, LinkedIn and Twitter). Social media will not be used for conversations, only for advertisement purposes. Postings will include only the information that is included on the print poster. Recruitment at clinics will be done via posters.

Participants will fill out clinical questionnaires (COMPASS31 and DePaul Symptom Questionnaire) and complete a cognitive function test using BrDI software developed by Dr. Lauren Sergio. This software program is located on a lab laptop and consists of trials whereby participants move a mouse on a screen in particular directions as instructed. They will then complete the following in random order: 1) breathe hypoxic gas (10% O2) for 5 minutes; 2) breathe hypercapnic gas (5% CO2) for 5 minutes; 3) breathe at a rate of 6 breaths per minute (paced deep breathing); and 4) 10 minutes upright tilt (70 degrees on a tilt-table). Each trial will be separated by 10 minutes of supine rest. Participants will also complete a voluntary walking test whereby the distance walked in 6 minutes will be measured as an index of aerobic fitness. All of these trials will be conducted in 336 Calumet College and will be conducted both before and after the 8-weeks of inspiratory muscle training described below (i.e. at both their first and second visits).

All participants will be equipped to measure heart rate, beat-to-beat blood pressure, brain blood flow, ventilation and end-tidal gases. Heart rate (HR) will be measured by electrocardiogram (ECG), and blood pressure will be monitored using a beat-by-beat non-invasive blood pressure device on the middle finger (NexFin). Brain blood flow velocity from the middle cerebral artery in the brain will be recorded using ultrasound and a 2MHz probe (Multigon Industries Inc.) positioned on the temple and held in place by an adjustable head-band. Respiratory outcomes such as ventilation, tidal volume, breathing frequency, exhaled gases will be measured through a mouthpiece that will be attached to a pneumotachometer (a nose plug will be worn).

These experiments will take approximately 2.5 hours per testing session.

Using commercially available devices, the 8-week inspiratory muscle training protocol consists of using 80% of maximal inspiratory pressure (determined in lab), 3x per week, 6 sets of 6 repetitions. Each set will be separated by decreasing lengths of time over the 8 weeks starting at a 30 second interim. This totals 36 inhalations 3 times per week. Progress will be determined via weekly phone calls with the participants and progress will also be logged by participants over the 8 weeks

ELIGIBILITY:
Inclusion Criteria:

* Control participants will be free of previously diagnosed cardiovascular, metabolic, autonomic, or respiratory disease.
* COVID-19 participants will have both an official diagnosis and an official clearance of COVID-19. Patients will have long-haul symptoms for at least 3 months. Patients will be recruited via media, social media and clinical collaborators.
* ME/CFS participants will be recruited via media, social media and clinical collaborators. Only those with mild to moderate symptoms who can complete a 6 minute walk test will be recruited.

Exclusion Criteria:

* severe symptoms of chronic fatigue syndrome
* inability to stand on a tilt table
* inability to walk for 6 minutes
* previous cardiorespiratory disease (except for COVID long-hauler symptoms and chronic fatigue syndrome itself)
* inability to understand and read English.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-05-09 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Chemoreflex function | 8 weeks
  Ventilatory responses to the administration of 10% hypoxia or 5% hypercapnia will be measured.
Clinical autonomic function | 8 weeks
  Cardiovascular responses to autonomic battery of tests
Vascular function | 8 weeks
  Brachial artery dilation response to 5 minutes of circulatory occlusion (flow-mediated dilation).
Cognitive function | 8 weeks
  Performance on proprietary cognitive function software

SECONDARY OUTCOMES:
Cardiorespiratory fitness | 8 weeks
  6-minute walk distance
ME symptoms | 8 weeks
  DePaul symptom questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Heather Edgell, PhD, Principal Investigator — York University
Locations (1):
- York University, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
No individual data will be shared with anyone unless legally required to do so.

REFERENCES:
- [Derived] Edgell H, Pereira TJ, Kerr K, Bray R, Tabassum F, Sergio L, Badhwar S. Inspiratory muscle training improves autonomic function in myalgic encephalomyelitis/chronic fatigue syndrome and post-acute sequelae of SARS-CoV-2: A pilot study. Respir Physiol Neurobiol. 2025 Jan;331:104360. doi: 10.1016/j.resp.2024.104360. Epub 2024 Oct 6. PMID 39374820